CLINICAL TRIAL: NCT00288340
Title: Quantifying Abnormalities in Cortical Activation Associated With Auditory Hallucinations Using Functional Magnetic Resonance Imaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 050978; NARSAD
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Hallucinations
Keywords: psychotic disorders; auditory hallucinations; brain structure; psychiatric disorder with auditory hallucinations (at least one every 20 minutes); schizophrenia/schizoaffective disorder without auditory hallucinations
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Hallucinations | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1,2 (Active Comparator)
  Interventions: Device: functional magnetic resonance imaging

INTERVENTIONS:
Device: functional magnetic resonance imaging

SUMMARY:
The goal of the project is to characterize abnormalities in brain structure and function related to schizophrenia. The investigators will use advanced magnetic resonance imaging (MRI) techniques to measure the degree and distribution of neuronal activity during specific cognitive tasks, alterations in neuronal connectivity, and how these are related to disease symptoms and treatment.

DETAILED DESCRIPTION:
The goal of the project is to characterize abnormalities in brain structure and function related to schizophrenia. We will use advanced magnetic resonance imaging (MRI) techniques to measure the degree and distribution of neuronal activity during specific cognitive tasks, alterations in neuronal connectivity, and how these are related to disease symptoms and treatment. We will focus on changes in brain structure and function associated with frequent auditory hallucinations, one of the most disabling manifestations of schizophrenia, and with neuroleptic treatment. In order to address these aims, we will study four groups of subjects:

1. patients who have frequent auditory hallucinations,
2. patients who are beginning a regimen of anti-psychotic medication,
3. patients who do not have frequent hallucinations and are not changing medication strategies, and
4. age-matched normal controls. Each group will contain 15 subjects for a total of 60.

ELIGIBILITY:
Inclusion Criteria:

Investigators will study subjects who:

* Are between the ages of 18 and 65.
* Meet diagnostic criteria for any psychiatric disorder with auditory hallucinations (at least one every 20 minutes) including schizophrenia/schizoaffective disorder OR schizophrenia/schizoaffective disorder without auditory hallucinations.
* Have been treated with an antipsychotic drug for hallucinations at least three months or are unmedicated
* Are willing to change their current antipsychotic medication if indicated
* Are able to provide written consent

Normal controls must :

* Be between the ages of 18 and 65
* Not meet the diagnostic criteria for schizophrenia or schizoaffective disorder or other psychiatric disorder involving hallucinations
* Not currently be treated with an antipsychotic drug
* Be able to provide written consent

Exclusion Criteria:

Subjects and normal controls will be excluded from participation if there is:

* Evidence of non-psychiatric, chronic central nervous system (CNS) disease (such as brain injury or neurological disease)
* Contraindication to MRI, including prior claustrophobic reaction and severe movement disorder
* A recent change in menstrual status other than recent changes in oral or implanted contraceptive use (for females)
* A positive pregnancy result (for females)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-01; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
characterize abnormalities in brain structure and function related to schizophrenia | two scans over a six month period

CONTACTS AND LOCATIONS:
Overall Officials: Adam Anderson, Ph.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States